CLINICAL TRIAL: NCT05523466
Title: Effect of Acupuncture on Heart Rate Variability in Individuals With Multiple Sclerosis
Brief Title: Effect of Acupuncture on Heart Rate Variability in Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Talita Dias da Silva, Clinical professor, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1239/2018
Record Dates: First submitted 2022-07-25; First posted 2022-08-31 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active-Sham group (Experimental): will start with 5 sessions (1 per week) of active acupuncture combined with HRV evaluation for 20 min. After a 2-week washout, this group will be reallocated to another 5 sessions (1 per week) of sham acupuncture for 20 min combined with HRV evaluation.
  Interventions: Other: Acupuncture Active; Other: Acupuncture Sham
- Sham-Active group (Experimental): will start an allocated 5 sessions (1 per week) of sham acupuncture combined with HRV evaluation, and after a 1-week washout period will be reallocated to 5 sessions (1 per week) of active acupuncture combined with HRV evaluation.
  Interventions: Other: Acupuncture Active; Other: Acupuncture Sham

INTERVENTIONS:
Other: Acupuncture Active — Immediately after the placement of the Polar V800, an instrument for analyzing heart rate variability, the placing of needles at the points carefully selected for this research begins. The needling will proceed for the Active acupuncture using specific Traditional Chinese Acupuncture points: E36, BP6, F3, IG4, for 20 minutes.
Other: Acupuncture Sham — Immediately after the placement of the Polar V800, an instrument for analyzing heart rate variability, the placing of needles at the points carefully selected for this research begins. The needling will proceed for the Sham acupuncture using sham points (points not recognized as Acupuncture points), with the duration of 20 minutes

SUMMARY:
The Objective of this study is to evaluate the heart rate variability in individuals with multiple sclerosis during the applicability of Acupuncture, to analyze the behavior of the autonomic nervous system before, during, and after therapy and the changes of the condition.

DETAILED DESCRIPTION:
A double-blinded randomized sham-controlled crossover trial with a 1:1 allocation ratio will be conducted, 40 individuals without previous illness will be evaluated, who will constitute the control group and 40 individuals with MS will constitute the experimental group, paired by age and gender. All participants will undertake active or sham acupuncture sessions. Active-Sham group will start with 5 sessions (1 per week) of active acupuncture combined with HRV evaluation for 20 min. After a 2-week washout, this group will be reallocated to another 5 sessions (1 per week) of sham acupuncture for 20 min combined with HRV evaluation. Meanwhile, Sham-Active group will carry out the opposite protocol, participants will start an allocated 5 sessions (1 per week) of sham acupuncture combined with HRV evaluation, and after a 1-week washout period will be reallocated to 5 sessions (1 per week) of active acupuncture combined with HRV evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with Multiple Sclerosis
* Aged over 18 years
* Motor and intellectual capacity to understand the evaluations
* Light and moderate functional classification levels (EDSS scale)
* Who accept to participate in the study through agreement with informed consent form

Exclusion Criteria:

* Do not understand the evaluations
* Cardiac diseases that impede the assessment of HRV
* Have a cardiac pacemaker.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Changes in the Heart Rate Variability after intervention | 84 days
  the capture strap will be placed on the volunteers' chests, and the heart rate receiver (V800, Polar) will be placed on their wrists

CONTACTS AND LOCATIONS:
Overall Officials: Celso Ferreira, Dr, Principal Investigator — Federal University of São Paulo

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2019-01-18): https://cdn.clinicaltrials.gov/large-docs/66/NCT05523466/Prot_000.pdf
  • Informed Consent Form (2019-01-18): https://cdn.clinicaltrials.gov/large-docs/66/NCT05523466/ICF_001.pdf